CLINICAL TRIAL: NCT00720252
Title: Can Ultrasound Replace Amniocentesis for Confirming Fetal Lung Maturation Among Premature Fetuses?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: TECHNICAL ISSUES
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0029-08-EMC
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Fetal Lung Maturity
MeSH Terms: interventions — Ultrasonography

ARMS (1):
- A (Experimental)
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — To measure intratracheal flow volume (and peak velocity) displaced during breathing cycle in premature fetuses.

SUMMARY:
The purpose of this study is to measure prenatally with ultrasound the intratracheal flow volume displaced during breathing cycle in premature fetuses and to check whether a relationship exists between the inspired fluid and fetal lung maturation.

ELIGIBILITY:
Inclusion Criteria:

* Women delivering between 27 to 37 weeks.
* Women undergoing amniocentesis for determining fetal lung maturity between 27 to 37 weeks.

Exclusion Criteria:

* Major fetal malformation.
* Oligohydramnios or rupture of membranes diagnosed before 24 weeks of gestation.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To check whether a threshold exists between peak velocity and/or volume of fluid inspired by the fetus and lung maturation. | end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. OB/GYN, HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] Kitterman JA. Fetal lung development. J Dev Physiol. 1984 Feb;6(1):67-82. No abstract available. PMID 6368667
- [Background] Kalache KD, Chaoui R, Bollmann R. Doppler assessment of tracheal and nasal fluid flow during fetal breathing movements: preliminary observations. Ultrasound Obstet Gynecol. 1997 Apr;9(4):257-61. doi: 10.1046/j.1469-0705.1997.09040257.x. PMID 9168577